CLINICAL TRIAL: NCT03860012
Title: Evaluating the Efficacy of Weekly Folic Acid in Pediatric Inflammatory Bowel Disease Patients on Methotrexate
Brief Title: Folic Acid in Pediatric Inflammatory Bowel Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Folic acid in Peds IBD
Record Dates: First submitted 2019-02-13; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: methotrexate; folic; acid
MeSH Terms: conditions — Inflammatory Bowel Diseases; Heartburn | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: All patients will receive 800mcg of supplemental folic acid per week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Folic Acid 800 mcg once weekly (Experimental): Patients on daily folic acid with a normal baseline folate level will be switched to once weekly dosing.
  Interventions: Drug: Folic Acid

INTERVENTIONS:
Drug: Folic Acid — Patients on daily folic acid with a normal baseline folate level will be switched to once weekly dosing.
  Other Names: Folate

SUMMARY:
Inflammatory bowel disease often requires immunomodulators, such as methotrexate, to maintain disease remission. This medication is administered as one dose weekly. Methotrexate can cause folic acid deficiency, so the current recommendation is to give daily folic acid supplementation while on methotrexate. Standard of care is to administer folic acid supplements daily. Patient compliance with daily folic acid is often suboptimal. The rationale is that weekly folic acid supplementation is as efficacious as daily dosing, and less frequent dosing likely will help improve patient compliance. The optimal dosing schedule of folate supplementation in relation to methotrexate is not known and there are not many research studies that have studied changing dosing of folate supplementation. One particular research study examined the effect of different dosing of folic acid supplements in patients with rheumatoid arthritis taking methotrexate. The study showed that folic acid at two different doses per week (5 mg low dose vs 27.5 mg high dose) did not effect the efficacy of methotrexate therapy, and patients who were on either folic acid supplementation had lower toxicity scores compared to patients not on folic acid supplementation. This study shows that folic acid dosed once per week can be useful in preventing methotrexate toxicity for rheumatoid arthritis patients. There were no studies that could be found that have studied this correlation for pediatric inflammatory bowel disease. Based on this current study, once weekly dosing of folic acid in IBD patients on methotrexate has the potential to be as efficacious as daily dosing.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of once weekly supplemental folic acid dosing compared to daily dosing in patients with inflammatory bowel disease (IBD) on methotrexate.

The study population is pediatric patients (ages 2-21) with inflammatory bowel disease on methotrexate who are receiving supplemental folic acid. The current standard of care is to administer folic acid supplements on a daily basis.

This will be a prospective study involving pediatric IBD patients on methotrexate. Each patient's baseline folate levels and other routine labs at enrollment (time zero) will function as their control at the conclusion of the study.

Doses will be standardized prior to study initiation. All patients will receive 800mcg of supplemental folic acid per week. IBD patients are typically evaluated and have lab draws every 6 months. For our study, labs will be obtained as routine labs (CBC, CMP) and a baseline folate level at the time of enrollment. Once these labs are obtained, patients with normal folate levels will qualify for inclusion in the study. They will be started on once weekly folate dosing. During the course of the study, if patients develop low folate levels, they will be removed from the study and placed back on daily doses of folate.

ELIGIBILITY:
Inclusion Criteria:

1. inflammatory bowel disease
2. on methotrexate at appropriate dosing
3. normal folate levels at onset of study
4. treatment with folic acid
5. ages 2-21 years

Exclusion Criteria:

1. abnormal folate levels
2. age > 21 or less than 2

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Folate level | at 6 months
  Evaluation of Folate level
Evaluation of Folate level | at 12 months
  Evaluation of Folate level

CONTACTS AND LOCATIONS:
Overall Officials: Tsega A Temtem, MD, Principal Investigator — UTHSC
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bermejo F, Algaba A, Guerra I, Chaparro M, De-La-Poza G, Valer P, Piqueras B, Bermejo A, Garcia-Alonso J, Perez MJ, Gisbert JP. Should we monitor vitamin B12 and folate levels in Crohn's disease patients? Scand J Gastroenterol. 2013 Nov;48(11):1272-7. doi: 10.3109/00365521.2013.836752. Epub 2013 Sep 25. PMID 24063425
- [Result] Bermejo F, Algaba A, Guerra I, Gisbert JP. Response to letter: folate deficiency in Crohn's disease. Scand J Gastroenterol. 2014 Feb;49(2):255-6. doi: 10.3109/00365521.2013.869829. Epub 2013 Dec 16. PMID 24328943
- [Result] Dhir V, Sandhu A, Kaur J, Pinto B, Kumar P, Kaur P, Gupta N, Sood A, Sharma A, Sharma S. Comparison of two different folic acid doses with methotrexate--a randomized controlled trial (FOLVARI Study). Arthritis Res Ther. 2015 Jun 11;17(1):156. doi: 10.1186/s13075-015-0668-4. PMID 26063325
- [Result] Dupont-Lucas C, Grandjean-Blanchet C, Leduc B, Tripcovici M, Larocque C, Gervais F, Jantchou P, Amre D, Deslandres C. Prevalence and Risk Factors for Symptoms of Methotrexate Intolerance in Pediatric Inflammatory Bowel Disease. Inflamm Bowel Dis. 2017 Feb;23(2):298-303. doi: 10.1097/MIB.0000000000001014. PMID 28107279
- [Result] Heyman MB, Garnett EA, Shaikh N, Huen K, Jose FA, Harmatz P, Winter HS, Baldassano RN, Cohen SA, Gold BD, Kirschner BS, Ferry GD, Stege E, Holland N. Folate concentrations in pediatric patients with newly diagnosed inflammatory bowel disease. Am J Clin Nutr. 2009 Feb;89(2):545-50. doi: 10.3945/ajcn.2008.26576. Epub 2008 Dec 30. PMID 19116333
- [Result] Kaskel FJ, Bamgbola OF. Validation of a composite scoring scheme in the diagnosis of folate deficiency in a pediatric and adolescent dialysis cohort. J Ren Nutr. 2008 Sep;18(5):430-9. doi: 10.1053/j.jrn.2008.05.009. PMID 18721738
- [Result] Pan Y, Liu Y, Guo H, Jabir MS, Liu X, Cui W, Li D. Associations between Folate and Vitamin B12 Levels and Inflammatory Bowel Disease: A Meta-Analysis. Nutrients. 2017 Apr 13;9(4):382. doi: 10.3390/nu9040382. PMID 28406440
- [Result] Park JA, Shin HY. Influence of genetic polymorphisms in the folate pathway on toxicity after high-dose methotrexate treatment in pediatric osteosarcoma. Blood Res. 2016 Mar;51(1):50-7. doi: 10.5045/br.2016.51.1.50. Epub 2016 Mar 25. PMID 27104192
- [Result] Scaglione F, Panzavolta G. Folate, folic acid and 5-methyltetrahydrofolate are not the same thing. Xenobiotica. 2014 May;44(5):480-8. doi: 10.3109/00498254.2013.845705. Epub 2014 Feb 4. PMID 24494987

DOCUMENTS (1):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03860012/Prot_000.pdf